CLINICAL TRIAL: NCT02945397
Title: Effect Evaluation of the Work Rehabilitation Effort "Best iLag"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Norwegian Labour and Welfare Administration Tromso (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Best iLag
Record Dates: First submitted 2016-09-30; First posted 2016-10-26 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Musculoskeletal Pain; Work Related Illnesses; Burnout, Professional
Keywords: Return to work; Work rehabilitation; Sick-leave
MeSH Terms: conditions — Musculoskeletal Pain; Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual activity (Active Comparator): The individual activity consists of a 3 month membership card at a given gym. This is in addition to regular follow-up from welfare authorities.
  Interventions: Behavioral: Individual activity
- Group-based activity (Active Comparator): The group-based activity consists of a 3 month group activity with weekly gatherings, focusing on coping, goal-setting and relevant information regarding available public services. This is in addition to regular follow-up from welfare authorities.
  Interventions: Behavioral: Group-based activity

INTERVENTIONS:
Behavioral: Group-based activity — Regular follow-up from welfare authority as well as a 3 month group activity with weekly gatherings, focusing on coping, goal-setting and relevant information regarding available public services.
  Arms: Group-based activity
Behavioral: Individual activity — Regular follow-up from welfare authority as well as a 3 month membership card at a given gym.
  Arms: Individual activity

SUMMARY:
The study compares the effect of a group-based activity with an individual work-out activity on work participation.

DETAILED DESCRIPTION:
The study is an RCT comparing the effect of a group-based intervention with an individual work-out intervention on work participation. The target group is persons who are at risk of leaving the work force due to health issues, and people currently outside the work force. The interventions have a time-span of 3 months. Survey data will be collected at baseline, after three months (after intervention has ended), and after 15 months. Survey data include information on lifestyle, self-reported health, subjective health complaints and readiness for work. Register data on employment and welfare benefits will be collected from two years in advance of inclusion, and five years after inclusion. According to power calculations, the study will need 322 participants.

In addition to the effect evaluation, a process evaluation will also be performed. The process evaluation will examine content quality and adherence to guidelines, as well as feasibility of the group intervention. The process evaluation will consist of some survey data as well as interviews with service providers and participants.

ELIGIBILITY:
Inclusion Criteria:

* Desire to work
* Understand Norwegian sufficiently to complete surveys

Exclusion Criteria:

* Not able to participate in the interventions due to personal or health-related constraints.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Number of days at work during follow-up period measured through data from the Norwegian Labour and Welfare Administration´s databases. | 7 years

SECONDARY OUTCOMES:
Subjective health complaints measured through questionnaire data. | 15 months
  Subjective health complaints inventory
Fatigue measured through questionnaire data. | 15 months
  Chalder fatigue questionnaire
Self-rated health measured through questionnaire data. | 15 months
  Global health question
Sleep measured through questionnaire data. | 15 months
  Sleep (single items)
Alcohol use measured through questionnaire data. | 15 months
  The Alcohol Use Disorders Identification Test
Quality of life measured through questionnaire data. | 15 months
  EQ-5D (Health-related quality of life + visual analogue scale)
Regular exercise measured through questionnaire data. | 15 months
  Regular exercise (single items)
Bullying measured through questionnaire data. | 15 months
  Bullying (single items)
Social support measured through questionnaire data. | 15 months
  Non-directive and Directive Support Survey
Coping measured through questionnaire data. | 15 months
  Theoretically Originated Measure of Cognitive Activation Theory of Stress
Work readiness measured through questionnaire data. | 15 months
  Readiness for Return to Work Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Torill Tveito, Principal Investigator — Uni Research Health
Locations (1):
- Uni Research, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No